CLINICAL TRIAL: NCT03130920
Title: Comparison of Hepatoprotective Effect From Ischemia-reperfusion Injury of Remote Ischemic Preconditioning of the Liver vs. Local Ischemic Preconditioning of the Liver During Human Liver Resections
Brief Title: Hepatoprotective Effect of Remote vs Local Preconditioning of Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Mislav Rakić, MD, Head of hepatobilliary Department of surgery, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHDubrava
Record Dates: First submitted 2017-04-01; First posted 2017-04-27 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Liver Metastases
Keywords: preconditioning, resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Remote ischemic preconditioning (Active Comparator)
  Interventions: Procedure: Preconditioning
- Local ischemic preconditioning (Active Comparator)
  Interventions: Procedure: Preconditioning

INTERVENTIONS:
Procedure: Preconditioning — Local ischemic preconditioning (LIPC) is process during which a short period of ischemia is followed by a period of reperfusion prior to the prolonged ischemia which seems to render organs more tolerant to the IR(ischemic-reperfusion) injury.
  Remote ischemic preconditioning (RIPC) involves the protection of an organ from prolonged ischemia by brief periods of ischemia and reperfusion to a remote organ.
  Arms: Local ischemic preconditioning; Remote ischemic preconditioning

SUMMARY:
The aim of this study is to evaluate hepatoprotective effect from ischemia-reperfusion injury of remote ischemic preconditioning of the liver against local ischemic preconditioning of the liver during human liver resections.

DETAILED DESCRIPTION:
In this randomized control study, a total of 60 patients were randomized into 3 groups: remote ischemic precondition group - RIPC (3 intervals of 5 minute right upper limb ischemia with 3 intervals of 5 minute reperfusion), local ischemic precondition group - LIPC (15 minutes of inflow liver occlusion followed by 10 minutes of reperfusion before liver transection), control group - CG (group without ischemic preconditioning before liver transection). Patients were also stratified according to the extent of the hepatectomy. Hepatoprotective effect was evaluated by comparing serum transaminase levels, bilirubin levels, albumin, and protein levels, coagulograms and pathohistological exams. We also measured flow rate by Doppler ultrasound of hepatic artery and portal vein before and after preconditioning.

ELIGIBILITY:
Inclusion Criteria:

* patients with colorectal cancer liver metastasis all of which signed an informed consent

Exclusion Criteria:

* having any other underlying liver disease, or preoperative increased liver transaminase, bilirubin
* patients with chronic cardiac, pulmonary or renal disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Change in synthetic liver function | Preoperatively, first, third and seventh postoperative day
  We measured residual synthetic liver function and liver ischemic-reperfusion injury by value level of bilirubin, total proteins, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), glutamic aminotransferase (ƴGT), cholinesterase, alkaline phosphatase (AP), coagulogram.

SECONDARY OUTCOMES:
Flow through the hepatic artery and portal vein | Before and after preconditioning
  During operation we preformed Doppler ultrasonography of hepatic artery and portal vein.
Liver histology evaluation | Up to 10 days after operation
  Liver paraffin-embedded, standard haematoxylin-eosin stained sections were analysed postoperatively to evaluate the ischemic reperfusion injury . According to Rodriguez et al. four elements of the liver histology were analysed: steatosis (micro vesicular and macro vesicular) in 4 grades, degree of sinusoidal congestion and dilatation in 3 grades, leukocyte infiltration in 3 grades and necrosis (focal, confluent, or zonal) in 3 grades.26 Each biopsy was evaluated by a single pathologist blinded to the treatment allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Patrlj, Study Chair — Clinical Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No